CLINICAL TRIAL: NCT07140952
Title: Fueling Strong Hearts for a Strong South Carolina
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clemson University (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25ISA1475971
Record Dates: First submitted 2025-08-21; First posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Stroke; Obesity &Amp; Overweight
Keywords: Lifestyle Management; Virtual Intervention
MeSH Terms: conditions — Stroke; Obesity; Overweight

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- StrongSC (Experimental): The Strong SC arm combines the StrongPeople StrongHearts program with a supplemental medically tailored grocery (MTG) program.
  Interventions: Behavioral: Strong SC
- StrongPeople StrongHearts (Experimental): The StrongPeople StrongHearts arm follows the standard 12-week StrongPeople StrongHearts group program, systematically adapted to the needs and abilities of community-dwelling, chronic stroke survivors.
  Interventions: Behavioral: StrongPeople StrongHearts
- Control (No Intervention): No intervention will be administered during the wait-list control period.

INTERVENTIONS:
Behavioral: Strong SC — The Strong SC intervention combines the StrongPeople StrongHearts program with a supplemental medically tailored grocery program. The StrongPeople StrongHearts program is a 12-week group program, with two meetings per week, that incorporates education on nutrition and physical activity for weight management and cardiovascular health, as well as strength training and aerobic exercises. The supplemental MTG program will utilize a grocery delivery platform(s) to deliver a weekly medically tailored grocery box of produce worth approximately $30 (costs covered by grant funds). Box contents will be tailored by the PI, who is a registered dietitian licensed in South Carolina, to participants' nutrition needs and functional abilities (e.g., pre-cut vegetables for participants with limited hand functionality). Participants will receive an allotment of produce each week, as well as a recipe(s) and virtual cooking demonstration providing practical strategies on incorporating each week's produce.
  Arms: StrongSC
Behavioral: StrongPeople StrongHearts — The StrongPeople StrongHearts program is a 12-week group program, with two meetings per week, that incorporates education on nutrition and physical activity for weight management and cardiovascular health, as well as strength training and aerobic exercises. Participants of this intervention will receive a systematically adapted version of this program tailored to the physical capacities of the target population (chronic stroke survivors). The systematically adapted version of StrongPeople StrongHearts will be used across both experimental arms in this study.
  Arms: StrongPeople StrongHearts

SUMMARY:
South Carolina is home to many survivors of stroke. After leaving the hospital and finishing therapies, stroke survivors often do not have the supports they need to fully recover. Many live with problems for a long time after their stroke, such as trouble walking or doing everyday tasks like cleaning, grocery shopping, or cooking. Research suggests that healthy habits, like moving more, eating well, and being at a healthy weight, can improve most of these disabilities. These habits can be hard to form alone though, especially in rural areas that may not have many healthy foods or places to exercise. Research-based programs can help people form healthy habits. These programs have not been tested in stroke survivors who have different needs though. The goal of this research project is to test StrongPeople StrongHearts, a health program, to see if it helps stroke survivors in South Carolina make better choices for their health and improve their quality of life. The program will be delivered online so that survivors in rural areas can be in the program. One group will also receive a weekly grocery box tailored to their needs to improve access to healthy foods. This study could help increase access to research-based programs for stroke survivors who do not have the supports they did soon after their stroke. This step is important for stroke survivors' long-term health and quality of life, the mission of the American Heart Association.

DETAILED DESCRIPTION:
This study will be conducted virtually throughout the Pee Dee and Low Country regions of South Carolina. The purpose of this project is to determine the extent to which Strong SC, an intervention combining StrongPeople StrongHearts with a supplemental medically tailored grocery (MTG) program, impacts lifestyle behaviors and health outcomes of community-dwelling chronic stroke survivors with obesity, compared to the conventional StrongPeople StrongHearts intervention. A total of 50 community-dwelling chronic stroke survivors with overweight or obesity will be randomly assigned to one of three groups: 1) StrongPeople StrongHearts + supplemental MTG program (Strong SC); 2) the conventional StrongPeople StrongHearts program (SPSH); or 3) a wait-list control (CON). SPSH participants will have access to the supplemental MTG program following completion of the 12-week intervention and 12-week follow-up period, and CON participants will be enrolled in the Strong SC intervention following the 12-week intervention and 12-week follow-up period. Anthropometric measures, physical activity, physical and psychosocial function, diet quality, and food security (Aim 1) outcome measures will be assessed prior to the intervention (baseline), at 12 weeks (post), and at 24 weeks (follow-up). The RE-AIM (Reach, Effectiveness, Adoption, Implementation, and Maintenance) and Framework for Reporting Adaptations and Modifications-Expanded (FRAME) frameworks will be utilized to evaluate implementation outcomes and systematic adaptations to StrongPeople StrongHearts (Aim 2). Any StrongPeople StrongHearts program adaptations required, systematically made, and documented will apply to both the Strong SC and SPSH intervention groups.

ELIGIBILITY:
Inclusion Criteria:

1. age 45-80 years;
2. a diagnosis of stroke at least 6 months prior;
3. BMI > 25 kg/m2;
4. ability to follow instructions, complete training, and to communicate exertion, pain, and distress;
5. access to computer or smart phone with internet to participate in a virtual intervention; and
6. provision of informed consent. Individuals who meet inclusion criteria must complete the Physical Activity Readiness Questionnaire (PARQ) and be cleared for participation by a study exercise physiologist

Exclusion Criteria:

1. unstable cardiac arrhythmias, hypertrophic cardiomyopathy, severe aortic stenosis, angina or dyspnea at rest or during ADL's;
2. Alzheimer's or other dementias;
3. life expectancy <1 yr;
4. history of DVT or pulmonary embolism within 6 months;
5. severe hypertension with systolic >200 mmHg and diastolic >110 mmHg at rest;
6. history of seizures or currently prescribed anti-seizure medications; or
7. current enrollment in a rehabilitation trial to enhance physical or psychosocial recovery

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-06-27 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Physical Activity | Baseline, post-intervention (12 weeks), and follow-up (24 weeks)
  Physical activity will be assessed objectively with accelerometers as well as subjectively with the International Physical Activity Questionnaire-Short form
Stroke Impact Scale 3.0 (SIS) | Baseline, post-intervention (12 weeks), and follow-up (24 weeks)
  Subjective Physical and Psychosocial Function
Diet Quality | Baseline, post-intervention (12 weeks), and follow-up (24 weeks)
  Diet quality will be assessed with the Healthy Eating Index-2020, calculated from two 24-hour recalls collected using the Automated Self-Administered 24-hour recall. Diet quality will also be assessed with the 26-item Dietary Screener Questionnaire (DSQ).

SECONDARY OUTCOMES:
Weight | Baseline, post-intervention (12 weeks), and follow-up (24 weeks)
  Weight will be self-reported but measured using clinical-grade scales provided to participants for the course of the intervention.
Food Security | Baseline, post-intervention (12 weeks), and follow-up (24 weeks)
  Household food security will be assessed with the Six-item Short Form of the Food Security survey module developed by the USDA Economic Research Service

CONTACTS AND LOCATIONS:
Locations (1):
- Pee Dee Research and Education Center, Florence, South Carolina, United States